CLINICAL TRIAL: NCT01289067
Title: Predicting Response to Platinum Chemotherapy in Metastatic Castration Resistant Prostate Ca(mCRPC)Using a Genomic Signature for "BRCAness": A Phase II Prospective Open Label Clinical Trial of Satraplatin in Men With mCRPC Who Have Progressed on Docetaxel
Brief Title: Utilizing A Genomic Sig for "BRCAness" to Eval the Efficacy of Satraplatin in Men With Met. Castration Resistant Prostate Ca
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: William K. Oh (Other)
Collaborators: Prostate Cancer Foundation (Other)
Responsible Party: Sponsor-Investigator, William K. Oh, Chief, Division of Hematology/Medical Oncology, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 10-1222; Prostate Cancer Foundation (Other: Prostate Cancer Foundation)
Record Dates: First submitted 2011-01-07; First posted 2011-02-03 (Estimated); Results first posted 2018-02-13 (Actual); Last update posted 2018-02-13 (Actual); Status verified 2018-01

CONDITIONS: Prostate Cancer
Keywords: Metastatic; Castration Resistant; Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Metastasis | interventions — satraplatin; amminedichloro(cyclohexylamine)platinum(II)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Satraplatin, Single Arm (Other)
  Interventions: Drug: Satraplatin

INTERVENTIONS:
Drug: Satraplatin — Satraplatin 80mg/m2 day 1-5 every 35 days Prednisone 5 mg twice daily every 35 days
  Other Names: JM-118

SUMMARY:
The purpose of the study is to test genes for BRCAness(BRCA[BReast CAncer] gene) Studying these genes could help predict which patients would benefit from treatment with satraplatin, a medication being used for subjects who have failed prior chemotherapy. All subjects will have a biopsy of metastatic lesions to measure BRCAness (a gene signature). This gene signature may be able to predict response to satraplatin and a tool will be developed to be able to screen patients likely to benefit from satraplatin. Subjects will all receive Satraplatin days 1-5 and Prednisone 5 mg twice daily every 35 days. Response rates will be evaluated every 2 cycles or approximately every 9 weeks. Patients will be considered responders if they have measurable disease meeting criteria for partial or complete response. PSA will be measured day one of each treatment cycle. Each treatment cycle is 35 days.

DETAILED DESCRIPTION:
We will be developing a genomic based signature of "BRCAness" based on literature of genomic signatures from women with breast cancer and germline BRCA mutations.The "BRCAness" breast cancer signature will differentiate germline BRCA 1/2 breast cancers from standard estrogen-receptor (+) breast cancers. We will obtain a library of genomic signatures Recently these techniques have been used to develop a transcriptional "signature" for androgen receptor (AR) activity in men with CRPC(Castration Resistant Prostate Cancer). The investigator will apply the "BRCAness" breast cancer signature to pathological prostate cancer specimens to determine the percentage of patients in the overall prostate cancer population that express this signature, as well as the clinical and histological phenotype of this population.

This novel prostate cancer "BRCAness" signature will be developed over a period of 4-6 months. This "BRCAness" signature has not previously been evaluated in prostate cancer patients and would be expected, based on known characteristics of BRCA mutant breast and ovarian cancers, to be more platinum-responsive. Relevant clinical data, including histology, grade, stage, size of residual tumor, recurrence, and survival, will be obtained from outpatient and inpatient charts to perform subsequent correlative studies.

All patients enrolled in the phase II clinical trial with satraplatin will have pre-treatment biopsies of metastatic sites. All of the specimens will be frozen, batched and stored as previously described. We anticipate that all patients will be enrolled 16 months from when the trial opens. When the last patient is enrolled in the trial and all of the metastatic biopsies have been collected, they will be shipped in bulk on dry ice to laboratory for RNA(ribonucleic acid) isolation, RNA quality assessment and processing, microarray hybridization, microarray data quality assessment, and "BRCAness" prostate cancer signature application. Frozen biopsies will be processed for microarray analysis using laser capture microdissection and RNA amplification using adaptations of previously published methods. The application of the prostate cancer BRCAness signature will take place over two months.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically confirmed adenocarcinoma of the prostate.
2. Radiographic evidence of metastatic disease (Bone scan, CT(Computerized Tomography) scan, or MRI(Magnetic Resonance Imaging) are acceptable) amenable to image-guided biopsy.
3. Castrate levels of testosterone (testosterone <50 ng/dL) on androgen deprivation therapy (ADT). LHRH(luteinizing hormone releasing hormone)agonist therapy must continue while on study unless patient has previously undergone an orchiectomy.
4. The patient must have discontinued antiandrogens (bicalutamide, flutamide or nilutamide) 30 days prior to baseline PSA.
5. Progression on at least one line of a prior docetaxel-based chemotherapy.
6. Patients must have adequate organ and marrow function as defined below:

   * Absolute neutrophil count >1,500/μl
   * Platelets >100,000/μl
   * GFR(glomerular Filtration Rate) >30 ml/min
   * ALT(Alanine transaminase) and AST(Aspartate transaminase) ≤ 2.5 X upper limit of normal (ULN) or ≤ 5 X ULN in patients with liver metastasis
7. Age > 18 years
8. Ability to take oral medications (pills must be swallowed whole)
9. ECOG (Eastern Cooperative Oncology Group) performance status 0-2
10. Ability to understand and the willingness to sign a written informed consent document
11. Patients must be willing to undergo an image-guided biopsy of a metastatic site on at least one occasion.
12. Patient agrees to utilize contraception while enrolled in the trial

Exclusion Criteria:

1. Patients who have received prior treatment with a platinum chemotherapy.
2. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection (requiring antifungal, antibiotic or antiviral therapy), history of symptomatic congestive heart failure (NYHC (New York Heart Association Classification) III), unstable angina pectoris, cardiac arrhythmia (uncontrolled SVT(Super ventricular tachycardia)or any VT(ventricular tachycardia), or psychiatric illness/social situations that would limit compliance with study requirements.
3. Patients with a medical contraindication to image-guided biopsies
4. Patients with a severe allergic reaction to satraplatin compounds.
5. Has a history of a prior malignancy with the exception of the following: adequately treated basal cell or squamous cell skin cancer, or other cancers for which the subject has been disease-free for at least 5 years.
6. Has had radiation therapy within 30 days prior to being registered for protocol therapy.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2010-12; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William K Oh, M.D., Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai Medical Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began in December 2010. Thirteen (13) patients from Mount Sinai Medical Center were enrolled to the study between January 27, 2011 and March 7, 2013.
Period: Overall Study
Arm/Group | Satraplatin, Single Arm
Started | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Satraplatin, Single Arm
Number analyzed (Participants) | 13
Age, Continuous [Median (Full Range); unit: years] | 69 [54 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 13
Metastasis site [Number; unit: participants]
  Bone only | 6
  Lymph Node only | 4
  Visceral only | 0
  Bone and Lymph Node | 1
  Bone and Visceral | 3
  Lymph Node and Visceral | 1
  Bone, Lymph Node, and Visceral | 2
Gleason Score [Number; unit: participants] — Gleason scores range from 2 to 10, with 2 representing the most well-differentiated tumors and 10 the least-differentiated tumors. Least-differentiated tumors typically have a worse prognosis.
  participants
    Gleason 7 | 4
    Gleason 8 | 5
    Gleason 9 | 4
PSA [Median (Full Range); unit: ng/ml] — pre-treatment PSA
  ng/ml | 71.67 [0.04 to 3057]

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of Satraplatin as Second Line Therapy in Men With CRCP
Description: Patients with good tolerance of treatment who have a 30% PSA decline from their pre-treatment level within 3 months of treatment initiation will be considered responders provided objective tumor measurements are stable or also demonstrate response.
Time Frame: 3 months
Measure: Number; unit: participants
Arm/Group | Satraplatin, Single Arm
Number analyzed (Participants) | 13
participants
  responders | 4
  non-responders | 6
  not evaluable for response | 3

2. Secondary Outcome: Number of Days to Maximum Decline in PSA
Description: Response rate - Maximum decline in PSA that occurs during treatment.
Time Frame: baseline and 3 months
Population: Only responders included
Measure: Median (Full Range); unit: days
Arm/Group | Satraplatin, Single Arm
Number analyzed (Participants) | 4
days | 165.5 [68 to 236]

3. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression Free Survival is measured from the time of the initiation of therapy until the first date that recurrent or progressive disease is objectively documented. Progression is a composite endpoint that can be based upon PSA, objective measures of disease, symptoms or death. Time to disease progression.
Time Frame: up to 2 years
Measure: Median (Full Range); unit: days
Arm/Group | Satraplatin, Single Arm
Number analyzed (Participants) | 13
days
  Responders | 206 [73 to 356]
  Nonresponders | 35 [31 to 41]

4. Secondary Outcome: Overall Survival
Description: Patients followed for a minimum of 24 months or until death. Patients and/or their family members will be contacted via telephone calls or certified letter.
Time Frame: 24 months
Measure: Median (Full Range); unit: days
Arm/Group | Satraplatin, Single Arm
Number analyzed (Participants) | 13
days
  Responders | 570 [184 to 717]
  Nonresponders | 486 [147 to 644]

ADVERSE EVENTS:
Arm/Group | Satraplatin, Single Arm
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 10/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Satraplatin, Single Arm (N=13)
Leukopenia (Blood and lymphatic system disorders) | 3
Neutropenia (Blood and lymphatic system disorders) | 1
Thromboscytopenia (Blood and lymphatic system disorders) | 1
Fatigue (General disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Dysphagia (General disorders) | 2
Diarrhea (Gastrointestinal disorders) | 1

LIMITATIONS AND CAVEATS:
limitation include low sample size

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes